CLINICAL TRIAL: NCT01088906
Title: Study of Pemetrexed Disodium Plus Cisplatin as First-line Therapy in Patients With Advanced Non-squamous Cell Lung Cancer: a Phase IIA Pharmacogenomic Trial
Brief Title: Study of Pemetrexed Plus Cisplatin as First-line Therapy in Patients With Advanced Non-squamous NSCLC
Acronym: Phalcis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No safety reasons. Low recruitment.
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP09-01Phalcis; 2009-011327-31 (EudraCT Number)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: Phalcis; BRCA1; RAP80; TS; First line; Non-squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 ARM (Experimental): pemetrexed 500 mg/m2 IV + cisplatin 75 mg/m2 every 21 days
  Interventions: Drug: Pemetrexed/Cisplatin

INTERVENTIONS:
Drug: Pemetrexed/Cisplatin — Pemetrexed 500 mg/m2 IV followed by cisplatin 75 mg/m2 IV every 21 days. A cycle is 21 day.
  Other Names: The Tradename of pemetrexed is Alimta

SUMMARY:
This is a study of pemetrexed disodium plus cisplatin as first-line therapy in patients with advanced non-squamous cell lung cancer. This is a phase IIA pharmacogenomic trial.

DETAILED DESCRIPTION:
This is a non-randomized, phase IIA pharmacogenomic, open label, uncontrolled, efficacy study in patients with advanced non-squamous cell lung cancer as a first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-squamous NSCLC, that is not amenable to curative treatment with surgery or radiation therapy. This population encompasses advanced stage patients with select stage IIIB (with pleural or pericardial effusion) or stage IV disease. Histologic or cytologic documentation of recurrence is required in patients who were previously completely resected and now have progressive disease.
* Tissue must be available to generate and apply the genomics predictor. If not obtained at the time of diagnosis, then subject must consent to another biopsy. If patient had prior radiation therapy, tissue biopsy for genomics analysis must be outside radiation field.
* At least one, non-radiated, measurable lesion by RECIST criteria.
* ECOG performance status of 0 or 1
* No prior chemotherapy, biologic or targeted therapy for any malignancy.
* Prior radiation therapy is permitted if ≥1 week since completion of radiation treatment. Radiation must be <25% of bone marrow reserve.
* Age greater than 18 years.
* No previous or concomitant malignancy in the past 5 years other than surgical management for carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin.
* No other serious medical or psychiatric illness.
* Signed informed consent.
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 7 days prior to or at the time of enrollment based on a serum pregnancy test. Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determined by the patient and their health care team, during the study and for 3 months following the last dose of study drug.
* Required laboratory data within two weeks of enrollment:

  1. ANC or AGC greater than 1500 per uL
  2. Platelets greater than 100,000 per uL
  3. Total bilirubin less than 1.5mg/dL
  4. Creatinine clearance greater than or equal to 45 ml/min.
  5. SGOT/SGPT less than or equal to 3x/ULN except in presence of known hepatic metastases in which it may be up to 5x ULN.

Exclusion Criteria:

* Patients with squamous cell NSCLC.
* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent administration of any other anti-tumor therapy.
* Inability to comply with protocol or study procedures.
* Active infection requiring IV antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Documented symptomatic or untreated central nervous system (CNS) metastases (except if adequately treated and stable for at least 2 weeks).
* Major surgery within 2 weeks of study or other serious concomitant systemic disorders that, in the opinion or the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Myocardial infarction having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia or cardiac failure not controlled by medications.
* Have peripheral neuropathy of CTCAE Grade 1 or higher
* Contraindications to corticosteroids.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Unwillingness to stop taking herbal supplements while on study.
* Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study entry and throughout study enrollment as the distribution of pemetrexed in this fluid space is not fully understood.
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination.
* Have prior known allergic/hypersensitivity reaction to any of the components of study treatment
* Inability to discontinue administration of aspirin at a dose greater than 1300 mg/day or other non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days for long-acting agents such as piroxicam).
* Female patients that is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Sánchez Torres, MD, Study Chair — Spanish Lung Cancer Group
Locations (8):
- Spain (8):
  - H. Clínica Benidorm, Benidorm, Alicante
  - H. General de Elche, Elche, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Insular de Gran Canarias, Las Palmas de Gran Canaria, Las Palmas
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - MD Anderson, Madrid
  - Hospital 12 de Octubre, Madrid
  - H. Morales Messeguer, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Lung Cancer Group website — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: start date: 20 January 2010 and ended at 19 February 2014.
Groups:
- Experimental: Pemetrexed Plus Cisplatin: Pemetrexed 500 mg/m2 IV + cisplatin 75 mg/m2 every 21 days
  Pemetrexed/Cisplatin: Pemetrexed 500 mg/m2 IV followed by cisplatin 75 mg/m2 IV every 21 days. A cycle is 21 day. Total: 6 cycles.
Period: Overall Study
Arm/Group | Experimental: Pemetrexed Plus Cisplatin
Started | 57
Completed | 52
Not Completed | 5
Not completed — Inclusion error | 1
Not completed — Did not receive study treatment | 3
Not completed — Missing data | 1

BASELINE CHARACTERISTICS:
Population: Patients stage IV non-squamous lung cancer that take at least 1 cycle of study medication. Intention-to-treat population.
Groups:
- EXPERIMENTAL ARM: Pemetrexed 500 mg/m2 IV + cisplatin 75 mg/m2 every 21 days
  Pemetrexed/Cisplatin: Pemetrexed 500 mg/m2 IV followed by cisplatin 75 mg/m2 IV every 21 days. A cycle is 21 day. Total: 6 cycles.
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 62 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 39
Region of Enrollment [Number; unit: participants]
  Spain | 52
Smoking status [Number; unit: participants]
  Never | 5
  Former | 31
  Smoker | 16
ECOG [Number; unit: participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity and physical ability
  GRADES:
  ECOG UK:Unknown ECOG 0: Fully active ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  participants
    ECOG 0 | 14
    ECOG 1 | 33
    ECOG UK | 5
Histology [Number; unit: participants]
  Adenocarcinoma | 51
  Large Cell Lung Carcinoma | 1
Treatment compliance [Number; unit: participants]
  Cycle 1 completed | 1
  Cycle 2 completed | 7
  Cycle 3 completed | 6
  Cycle 4 completed | 8
  Cycle 5 completed | 4
  Cycle 6 completed | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of patients who have experienced a tumor response since the start of treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From start of treatment to end of follow up, up to 24 months
Population: The percentage of patients who have experienced tumor regression since the start of treatment (Complete response + Partial response) among the total of patients ORR = 26%
Measure: Number; unit: percentage of participants
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
percentage of participants
  Stable disease | 44
  Partial response | 22
  Complete response | 4
  Progression | 30
Statistical Analysis 1: Comparison: EXPERIMENTAL ARM; Test type: Superiority; p = 0.05, Regression, Logistic; Odds Ratio (OR) = 34

2. Secondary Outcome: Overall Survival
Description: Overall survival is measured from the date of enrollment to the date of death from any cause
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month | 11.267 [9.141 to 13.392]

3. Secondary Outcome: Time to Progression
Description: This interval is measured in months from the date of entry into the study until the first date of the appearance of new metastatic lesions or objective progression of the disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month | 5.633 [4.180 to 7.087]

4. Secondary Outcome: Time to Progression of Patients According the Results of Biomarker BRCA1
Description: This interval is measured from the date of entry into the study until the first date of the appearance of new metastatic lesions or objective progression of the disease for patients with biomarker BRCA1.
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The number of subjects analyzed depends on BRCA results
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  BRCA1 negative: number analyzed (Participants) | 26
  BRCA1 negative | 5.270 [3.443 to 7.097]
  BRCA1 positive: number analyzed (Participants) | 26
  BRCA1 positive | 3.430 [0.564 to 6.296]
  All patients (BRCA1 positive+negative) | 5.270 [2.678 to 7.862]

5. Secondary Outcome: Time to Progression of Patients According the Results of Biomarker RAP80
Description: This interval is measured from the date of entry into the study until the first date of the appearance of new metastatic lesions or objective progression of the disease.
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The subjects analyzed depends on RAP80 results.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  RAP80 negative: number analyzed (Participants) | 26
  RAP80 negative | 5.630 [2.416 to 8.844]
  RAP80 positive: number analyzed (Participants) | 26
  RAP80 positive | 3.430 [0.0 to 7.354]
  All patients (RAP80 positive+negative) | 5.370 [2.430 to 8.310]

6. Secondary Outcome: Time to Progression of Patients According the Results of Biomarker TS
Description: as for outcome 5
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The subjects analyzed depends on TS results.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  TS negative: number analyzed (Participants) | 26
  TS negative | 5.630 [0.249 to 11.011]
  TS positive: number analyzed (Participants) | 26
  TS positive | 3.330 [2.590 to 4.070]
  All patients (TS positive+negative) | 3.430 [1.738 to 5.122]

7. Secondary Outcome: Overall Survival of Patients According the Results of Biomarker BRCA1
Description: Overall survival is measured from the date of enrollment to the date of death from any cause
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The subjects analyzed depends on BRCA1 results.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  BRCA1 negative: number analyzed (Participants) | 26
  BRCA1 negative | 12.270 [7.605 to 16.935]
  BRCA1 positive: number analyzed (Participants) | 26
  BRCA1 positive | 8.400 [0.864 to 15.936]
  All patients (BRCA1 positive+negative) | 10.570 [6.921 to 14.219]

8. Secondary Outcome: Overall Survival of Patients According the Results of Biomarker RAP80
Description: Overall survival is measured from the date of enrollment to the date of death from any cause
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The subjects analyzed depends on RAP80 results.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  RAP80 negative: number analyzed (Participants) | 26
  RAP80 negative | 10.570 [0.00 to 24.843]
  RAP80 positive: number analyzed (Participants) | 26
  RAP80 positive | 9.600 [4.787 to 14.413]
  All patients (RAP80 positive+negative) | 10.570 [5.865 to 15.275]

9. Secondary Outcome: Overall Survival of Patients According the Results of Biomarker TS
Description: Overall survival is measured from the date of enrollment to the date of death from any cause.
Time Frame: From the date of enrollment until end of follow up, up to 24 months.
Population: The subjects analyzed depends on TS results.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | EXPERIMENTAL ARM
Number analyzed (Participants) | 52
Month
  TS negative: number analyzed (Participants) | 26
  TS negative | 12.270 [2.136 to 22.404]
  TS positive: number analyzed (Participants) | 26
  TS positive | 8.400 [0.473 to 16.327]
  All patients (TS positive+negative) | 11.270 [5.351 to 17.189]

ADVERSE EVENTS:
Time Frame: 25 months
Groups:
- Experimental Arm: Pemetrexed Plus Cisplatin: Pemetrexed 500 mg/m2 IV + cisplatin 75 mg/m2 every 21 days
  Pemetrexed/Cisplatin: Pemetrexed 500 mg/m2 IV followed by cisplatin 75 mg/m2 IV every 21 days. A cycle is 21 day. Total: 6 cycles.
Arm/Group | Experimental Arm: Pemetrexed Plus Cisplatin
All-Cause Mortality (participants affected / at risk) | 9/52
Serious Adverse Events (participants affected / at risk) | 25/52
Other Adverse Events (participants affected / at risk) | 40/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm: Pemetrexed Plus Cisplatin (N=52)
Lower member embolism (Vascular disorders) | 1 (1)
Stroke ischemic and pneumonia (Vascular disorders) | 1 (1)
Acute ischemia of lower limbs (Vascular disorders) | 1 (1)
Pulmonary thromboembolism (Vascular disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (5)
Disorientation and loss motor control (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyporexia (General disorders) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anorexy (General disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Impaired function renal (Renal and urinary disorders) | 2 (2)
Urinary infection (Renal and urinary disorders) | 1 (1)
General stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Oliguria (Endocrine disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Bilateral bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm: Pemetrexed Plus Cisplatin (N=52)
Hypersensitivity (Immune system disorders) | 1 (1)
Haemoglobin (Blood and lymphatic system disorders) | 40 (40)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 (20)
Neutrophils (Blood and lymphatic system disorders) | 14 (14)
Platelets (Blood and lymphatic system disorders) | 6 (6)
Edema (General disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neurotoxicity sensitive (Nervous system disorders) | 8 (8)
Conjunctivitis (Eye disorders) | 3 (3)
Fatigue (General disorders) | 35 (35)
Fever (General disorders) | 1 (1)
Ototoxicity (Ear and labyrinth disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dysgeusia (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 13 (13)
Mucositis (Gastrointestinal disorders) | 12 (12)
Nausea-vomiting (Gastrointestinal disorders) | 40 (40)
Impaired function renal (Renal and urinary disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Increase AST/ALT (Endocrine disorders) | 7 (7)
Hyporexia (Metabolism and nutrition disorders) | 7 (7)
Increase GGT (Metabolism and nutrition disorders) | 8 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
LDH increase (Metabolism and nutrition disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
26 February 2014: This study had a premature discontinuation due to the low recruitment rate of the study, not for safety reasons of the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No